CLINICAL TRIAL: NCT00801229
Title: The Effects of Vyvanse on the Driving Performance of Young Adults With ADHD: A Randomized, Double-Blind, Placebo-Controlled Study
Brief Title: Effect of Vyvanse on Driving in Young Adults With ADHD
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Collaborators: Shire (Industry)
Responsible Party: Principal Investigator, Joseph Biederman, MD, Chief of the Clinical and Research Programs in Pediatric Psychopharmacology and Adult ADHD, Massachusetts General Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2008P000971
Record Dates: First submitted 2008-12-02; First posted 2008-12-03 (Estimated); Results first posted 2011-08-25 (Estimated); Last update posted 2014-03-10 (Estimated); Status verified 2014-02

CONDITIONS: Attention Deficit/Hyperactivity Disorder(ADHD)
Keywords: ADHD; young adults; driving; Vyvanse; lisdexamfetamine
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity | interventions — Lisdexamfetamine Dimesylate

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Vyvanse (Active Comparator): Patients may be randomized to the active comparator arm. Participants randomized to this arm will receive 30, 50, or 70mg Vyvanse daily.
  Interventions: Drug: Vyvanse
- Placebo (Placebo Comparator): Patients may be randomized to the placebo comparator arm. Those randomized to this arm will receive 30, 50, or 70mg placebo daily.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Vyvanse — Vyvanse 30, 50, or 70 mg daily
  Other Names: Lisdexamfetamine
  Arms: Vyvanse
Drug: Placebo — Placebo 30, 50, 70 mg daily
  Arms: Placebo

SUMMARY:
The primary objective of the study is to assess the benefice of Vyvanse on the factors that cause impairments in driving behavior in individuals with ADHD using a driving simulation aimed at examining the factors that cause impairments in driving behavior in individuals with ADHD such as driving speed, collision risk, and visual attention of 60 young drivers (ages 18-24) with ADHD. We hypothesize: 1.) young adults with ADHD treated with Vyvanse will show lower velocity (speed) scores and spend less time driving over the posted speed limit in the driving simulation when compared to subjects taking a placebo; 2.) young adults with ADHD treated with Vyvanse will show a lesser likelihood to collide with a suddenly appearing peripheral object, less difficulty maintaining the vehicle within their lane, and a lesser likelihood of driving through stop signs and solid red traffic lights without slowing down when compared to subjects taking a placebo; and 3.) young adults with ADHD treated with Vyvanse will exhibit more focused visual attention on details in the visual field when compared to subjects taking a placebo while driving. In addition, young adults with ADHD treated with Vyvanse will exhibit less visual tunneling and shorter off-road glances when compared to subjects taking a placebo.

ELIGIBILITY:
Inclusion Criteria:

* Male and female outpatients, aged 18-24 years.
* Subjects meeting full criteria for the diagnosis of DSM-IV Attention Deficit Hyperactivity Disorder (ADHD), with onset of symptoms in childhood and persistence of impairing symptoms into adulthood as determined by clinical evaluation and/or ADHD module of structured diagnostic interview, completed by the study clinician.
* Absence of pharmacological treatment for ADHD for the past month.

Exclusion Criteria:

* Any other current psychiatric or medical condition determined to be clinically significant.
* Current use of psychotropics or any medication with clinically significant CNS effects.
* Individuals who have never held a valid driver's license.
* Mental retardation (IQ < 80).
* Individuals with a history of substance dependence or abuse within the past 6 months. Pregnant or nursing females.
* Known hypersensitivity to Vyvanse or amphetamines.
* Subjects with pre-existing structural cardiac abnormalities.
* Clinically significant abnormal screening values including:
* Laboratory values determined to be clinically significant.
* Consistent readings of hypertension (>140/90) during screening period (including screening and baseline visits), defined as two or more readings (each being the average of three measurements) at a single visit with systolic blood pressure, SBP > 140 and/or diastolic blood pressure, DBP, > 90, and confirmed by manual reading.
* Subjects with isolated incidences (of triplicate average BP) of SBP > 140 and/or DBP > 90 at baseline/week 0 visit, confirmed by manual reading, which are determined to be clinically significant.

Subjects with a clinically significant abnormality according to cardiology consultation (ECGs with clinically concerning intervals including PR, QTC, QRS, will be reviewed by cardiology).

Ages: 18 Years to 24 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 75 (Actual)
Dates: Start 2008-12; Primary Completion 2010-07 (Actual); Study Completion 2010-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Joseph Biederman, MD, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital, Cambridge, Massachusetts, United States

REFERENCES:
- [Derived] Biederman J, Fried R, Hammerness P, Surman C, Mehler B, Petty CR, Faraone SV, Miller C, Bourgeois M, Meller B, Godfrey KM, Baer L, Reimer B. The effects of lisdexamfetamine dimesylate on driving behaviors in young adults with ADHD assessed with the Manchester driving behavior questionnaire. J Adolesc Health. 2012 Dec;51(6):601-7. doi: 10.1016/j.jadohealth.2012.03.005. Epub 2012 Apr 20. PMID 23174471

RESULTS

PARTICIPANT FLOW:
Period: Signed Consent
Arm/Group | Vyvanse | Placebo
Started | 38 | 37
Completed | 35 | 34
Not Completed | 3 | 3
Not completed — Withdrawal by Subject | 2 | 2
Not completed — Found Ineligible | 1 | 1
Period: Received Study Drug/Placebo
Arm/Group | Vyvanse | Placebo
Started | 35 | 34
Completed | 31 | 30
Not Completed | 4 | 4
Not completed — Elevated SGOT level | 1 | 0
Not completed — Sub-threshold ADHD | 0 | 1
Not completed — Simulator sickness | 1 | 1
Not completed — Withdrawal by Subject | 1 | 0
Not completed — Lost to Follow-up | 0 | 1
Not completed — Adverse Event | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Vyvanse | Placebo | Total
Number analyzed (Participants) | 35 | 34 | 69
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 35 | 34 | 69
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: Years] | 22.26 (2.12) | 22.15 (1.99) | 22.20 (2.04)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14 | 16 | 30
  Male | 21 | 18 | 39
Region of Enrollment [Number; unit: participants]
  United States | 35 | 34 | 69

OUTCOME MEASURES:

1. Primary Outcome: Participants Experiencing Collisions During "Surprise Events" in Driving Simulator
Description: Initial results from a one hour driving simulation in the MIT AgeLab Driving Simulator as compared to second session in the simulator following a 6-week trial on Lisdexamfetamine or placebo. During the simulation, "surprise events," designed to test the participant's attention and driving, occurred. This outcome presents the difference in number of collisions experience by individuals treated with Vyvanse or Placebo.
Time Frame: 6 weeks
Population: Participants who completed the protocol, including endpoint Driving Simulation assessment, were analyzed (61 in total).
Measure: Number; unit: participants
Arm/Group | Vyvanse | Placebo
Number analyzed (Participants) | 31 | 30
participants | 8 | 17

ADVERSE EVENTS:
Arm/Group | Vyvanse | Placebo
Serious Adverse Events (participants affected / at risk) | 0/35 | 0/34
Other Adverse Events (participants affected / at risk) | 30/35 | 20/34
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Vyvanse (N=35) | Placebo (N=34)
Decreased Appetite (Metabolism and nutrition disorders) | 19 | 2
Mucosal Dryness (General disorders) | 9 | 1
Tense/Jittery (General disorders) | 8 | 2
Insomnia (General disorders) | 7 | 1
Headaches (General disorders) | 5 | 1
Gastrointestinal (Gastrointestinal disorders) | 3 | 2
Cold/Infection/Allergy (Infections and infestations) | 3 | 5
Agitated/Irritable (Psychiatric disorders) | 2 | 0
Sad/Down (Psychiatric disorders) | 2 | 0
Autonomic (General disorders) | 2 | 0
Musculoskeletal (Musculoskeletal and connective tissue disorders) | 2 | 4
Genitourinary (Renal and urinary disorders) | 2 | 0
Increased Energy (General disorders) | 1 | 0
Cardiovascular (Cardiac disorders) | 1 | 1
Decreased Energy (General disorders) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No